CLINICAL TRIAL: NCT04509492
Title: Role of EUS in Detection of Liver Metastasis Not Seen by CT or MRI During Staging of Pancreatic, Gastrointestinal, and Thoracic Malignancies.
Brief Title: Role of EUS in Detection of Liver Metastasis
Status: Completed | Type: Observational
Sponsor: Mahmoud Wahba (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Wahba, lecturer of medicine division of gastroenterology, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Ethical comittee N91/2020
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Liver Metastases; Pancreatic Neoplasms
Keywords: EUS; occult metastases
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endosonography; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound ( EUS ) — - EUS will be done to all patients. During EUS examination the liver will be examined thoroughly to detect hepatic focal lesions with possible EUS-FNA of any detected lesions.
  All EUS examination will being done by EUS linear array Echoendoscope, Pentax EG-3870UTK attached to Hitachi Avius US machine under Propofol deep sedation
  Other Names: EUS-FNA ( fine needle aspiration )

SUMMARY:
Liver metastasis may not be detected by CT and MRI due to their small size while they can be detected by EUS. Also, EUS-FNA has a great impact in improving the diagnostic accuracy of EUS. Objectives: To assess the feasibility of EUS in the detection of occult small hepatic focal lesions at the time of primary tumor staging, not seen by CT or MRI.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) was used firstly in 1980s as a diagnostic imaging technique for pancreatic lesions. It has the ability to detect the histological layers of the gastrointestinal (GI) tract wall as well as the periluminal structures.

EUS has been used to perform FNA from lesions that are difficult to access by conventional methods. EUS has the advantage of using both ultrasound and endoscopy to give the exact diagnostic features of the GI tract. The use of EUS was not limited to visualization only, but also in obtaining tissue biopsy for diagnostic purpose through EUS guided fine needle aspiration (FNA), and it has played a major role in revolutionizing the diagnosis of focal hepatic lesions as it is a minimally invasive procedure.

Abdominal imaging [CT, magnetic resonance imaging (MRI), and transabdominal ultrasonography (USG)] are the diagnostic tests of choice to detect hepatic lesions suspicious of metastasis.Unfortunately, these modalities are limited in their ability to detect hepatic lesions less than 1 cm.

In addition, although rare, percutaneous FNA for suspected metastatic lesions carries the risk of implantation metastasis. Although unable to completely visualize the entirety of the liver, EUS can detect small hepatic lesions that may be otherwise missed by conventional imaging. EUS can delineate detailed anatomy of the liver from the trans-gastric and trans-duodenal routes with the exception of the right posterior segments.

The prospect to obtain precise, ultrasound-guided biopsies of possible metastatic liver lesions can drastically alter the therapeutic conduct.

This, combined with limited adverse events, makes EUS an excellent modality to allow staging in malignant conditions. Due to the vicinity of the transducer to the liver, EUS provides detailed images of the liver segments and its vascular structures.

Based on the premise that EUS is more sensitive for the detection of small hepatic lesions then CT/MRI, Singh et al. proved that EUS was superior to CT scan (98% vs 92%, respectively) in diagnostic accuracy in its ability to detect the number of metastatic lesions in the liver and correctly diagnose the nature of the lesions .(Singh P etal.,2009) Endoscopic ultrasonography (EUS) has become an indispensable method for diagnosis and therapeutic procedures in gastroenterology and as experience with this technique is growing, new indications for EUS continue to emerge.

(Saraireh HA .,2017) Furthermore, the use of on-site cytopathology interpretation has further improved the diagnostic yield of EUS-FNA by helping to ensure that the samples obtained are representative of the target organ and adequate for diagnostic purposes.

Objectives: To assess the feasibility of EUS in detection of occult small hepatic focal lesions at the time of primary tumor staging, not seen by CT or MRI

All the patients will be subjected to:

1. Thorough history talking including;

   * Age
   * Sex
   * Comorbidity
2. Clinical general and local abdominal examination
3. Abdominal US & CT abdomen
4. laboratory investigations:

   1. complete blood count (CBC)
   2. Prothombin time ,INR
   3. Ceatinine , Urea
   4. Albumin
   5. ALT , AST
5. Virological test for HIV, HCV and HBV
6. CA-19-9 and alfa fetoproteins.
7. EUS will be done to all patients. During EUS examination the liver will be examined thoroughly to detect hepatic focal lesions with possible EUS-FNA of any detected lesions.

All EUS examination with be done by EUS linear array Echoendoscope, Pentax EG-3870UTK attached to Hitachi Avius US machine under Propofol deep sedation.

The collected data will be organized and statistically analyzed.

Data collection tool:

Data including study design, participant demographics, stage and type of pancreatic and GI malignancy will be extracted and recorded on electronic data collection sheet. Data will be pooled for various arms in trials: Individual data for each outcome were entered into the Comprehensive analysis. Pooled effects with 95%CI will be reported. Data will be analyzed separately for each arm.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with either pancreatic or gastrointestinal tumors and have undergone a CT scan of the abdomen with contrast or MRI before being referred for EUS for staging

Exclusion Criteria:

* Patients are younger than 12 years. Patients who previously known to have HCC. Patient unfit for deep sedation by Propofol injection. Patients with bleeding disorders contraindicating EUS-FNA

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 400 pt , both male and female above 12 years All patients diagnosed with either pancreatic or gastrointestinal tumors and have undergone a CT scan of the abdomen with contrast or MRI before being referred for EUS for staging
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
The number of patients with occult hepatic metastasis missed by CT or MRI during staging of pancreatic and GI malignancy. | 6 months
  pre-operative assessment of pancreatic neoplasms includes EUS examination to assess operability depending on the size, relation to blood vessels and metastasis. sometimes we found liver metastases missed during imaging evaluation by MRI and CT that could change the whole plan, so we aimed to study how frequent occult liver metastasis with be discovered during EUS staging of pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: hussein Okasha, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhatia V, Hijioka S, Hara K, Mizuno N, Imaoka H, Yamao K. Endoscopic ultrasound description of liver segmentation and anatomy. Dig Endosc. 2014 May;26(3):482-90. doi: 10.1111/den.12216. Epub 2013 Dec 19. PMID 24355092
- [Background] Prachayakul V, Aswakul P, Kachintorn U. EUS guided fine needle aspiration cytology of liver nodules suspicious for malignancy: yields, complications and impact on management. J Med Assoc Thai. 2012 Feb;95 Suppl 2:S56-60. PMID 22574530
- [Background] Saraireh HA, Bilal M, Singh S. Role of endoscopic ultrasound in liver disease: Where do we stand in 2017? World J Hepatol. 2017 Aug 28;9(24):1013-1021. doi: 10.4254/wjh.v9.i24.1013. PMID 28932347
- [Background] Eloubeidi MA, Khan AS, Luz LP, Linder A, Moreira DM, Crowe DR, Eltoum IA. Combined use of EUS-guided FNA and immunocytochemical stains discloses metastatic and unusual diseases in the evaluation of mediastinal lymphadenopathy of unknown etiology. Ann Thorac Med. 2012 Apr;7(2):84-91. doi: 10.4103/1817-1737.94527. PMID 22558013
- [Result] Wong JYY, Kongkam P, Ho KY. Training in endoscopic ultrasonography: An Asian perspective. Dig Endosc. 2017 May;29(4):512-516. doi: 10.1111/den.12802. Epub 2017 Feb 8. PMID 28066947
- [Result] Kim E, Telford JJ. Advances in endoscopic ultrasound, part 2: Therapy. Can J Gastroenterol. 2009 Oct;23(10):691-8. doi: 10.1155/2009/786212. No abstract available. PMID 19826645
- [Result] Srinivasan I, Tang SJ, Vilmann AS, Menachery J, Vilmann P. Hepatic applications of endoscopic ultrasound: Current status and future directions. World J Gastroenterol. 2015 Nov 28;21(44):12544-57. doi: 10.3748/wjg.v21.i44.12544. PMID 26640331